CLINICAL TRIAL: NCT03268941
Title: A 2-Part, Randomized, Double Blind and Open-Label, Placebo and Active-Comparator Controlled Trial to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics for TAK-906 in Subjects With Diabetes Mellitus and Gastroparesis or With Idiopathic Gastroparesis
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics (PK) and Pharmacodynamics (PD) for TAK-906 in Participants With Diabetes Mellitus and Gastroparesis (DG) or With Idiopathic Gastroparesis (IG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: TAK-906-1002; U1111-1196-9143 (Registry Identifier: WHO)
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Results first posted 2019-07-23 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus and Gastroparesis, Idiopathic Gastroparesis
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus; Gastroparesis | interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study has two parts: Part 1 (double-blind) and Part 2 (open-label).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1: Placebo (Placebo Comparator): TAK-906 placebo-matching (4x0 mg), capsule, orally, twice daily (BID) on Days 1-8 and once on Day 9 under fasted conditions.
  Interventions: Drug: TAK-906 Maleate Placebo
- Part 1: TAK 906 Maleate 5 mg (Experimental): TAK-906 maleate 1x5 mg, capsule, orally, BID and TAK-906 maleate placebo-matching (3x0 mg), capsules, orally, BID on Days 1-8, followed by TAK-906 maleate 1x5 mg, capsule, orally once on Day 9 under fasted conditions.
  Interventions: Drug: TAK-906 Maleate
- Part 1: TAK 906 Maleate 25 mg (Experimental): TAK-906 maleate 1x25 mg, capsule, orally, BID and TAK-906 maleate placebo-matching (3x0 mg), capsules, orally, BID on Days 1-8 followed by TAK-906 maleate 1x25 mg, capsule, orally, once on Day 9 under fasted conditions.
  Interventions: Drug: TAK-906 Maleate
- Part 1: TAK 906 Maleate 100 mg (Experimental): TAK-906 maleate 100 mg (4x25 mg), capsules, orally, BID on Days 1-8 and once a day on Day 9 under fasted conditions.
  Interventions: Drug: TAK-906 Maleate
- Part 2: TAK-906 Maleate 25 mg Fed Condition (Experimental): TAK-906 maleate 1x25 mg, capsule, orally, once on Day 1 of Period 1 under fed conditions (high fat breakfast), followed by a minimum 7- day washout.
  Interventions: Drug: TAK-906 Maleate
- Part 2: TAK-906 Maleate 25 mg Fasted Condition (Experimental): TAK-906 maleate 1x25 mg, capsule, orally, once on Day 1 of Period 2 under fasted conditions.
  Interventions: Drug: TAK-906 Maleate
- Part 2: Metoclopramide 10 mg (Active Comparator): Metaclopramide 10 mg, tablet, orally, once, 1 hour prior to breakfast on Day 1 in Part 2.
  Interventions: Drug: Metaclopramide

INTERVENTIONS:
Drug: TAK-906 Maleate — TAK-906 Maleate Capsules
  Arms: Part 1: TAK 906 Maleate 100 mg; Part 1: TAK 906 Maleate 25 mg; Part 1: TAK 906 Maleate 5 mg; Part 2: TAK-906 Maleate 25 mg Fasted Condition; Part 2: TAK-906 Maleate 25 mg Fed Condition
Drug: Metaclopramide — Metaclopramide Tablets
  Arms: Part 2: Metoclopramide 10 mg
Drug: TAK-906 Maleate Placebo — TAK-906 placebo-matching Capsules
  Arms: Part 1: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, PK and PD of TAK-906 in participants with Gastroparesis (GP).

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-906 maleate. TAK-906 maleate is being tested to treat people who have DG or IG. This study will assess the safety, tolerability, PK/PD and food effect of TAK-906 and will determine the effect of TAK-906 on gastric emptying (GE).

The study enrolled a total of 51 participants. This study will be conducted in two parts: Part 1 and Part 2. Part 1 will consist of 48 participants enrolled in 3 active treatment groups and 1 placebo group. Participants in Part 1 will be randomly assigned (by chance, like flipping a coin) to one of the 3 active treatment groups or 1 placebo group-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* TAK 906 maleate 5 mg
* TAK 906 maleate 25 mg
* TAK 906 maleate 100 mg
* Placebo

All participants who will complete Part 1 of the study will be eligible for enrollment in Part 2. Part 2 consisted of 21 participants who completed Part 1 and were assigned to the 2 open-label treatment groups as follow:

* TAK-906 maleate 25 mg Fed + TAK-906 maleate 25 mg Fasted: crossover design, with a minimum 7-day washout in doses of each period.
* Metoclopramide 10 mg

This multi-center trial will be conducted the United States. The overall time to participate in this study is approximately 8 weeks. Participants will make a final visit to the clinic 10-14 days after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible for participation in this trial, the participant must:

1. Has a documented diagnosis of diabetes mellitus gastroparesis (DG) or idiopathic gastroparesis (IG).
2. Has a body mass index (BMI) greater than or equal to (>=) 18 and less than or equal to (<=) 40 kilogram per square meter (kg/m^2) at the Screening Visit.
3. Be a non-smoker who has not used tobacco or nicotine-containing products (example, nicotine patch) for at least 6 months prior to trial drug administration of the initial dose of trial drug/invasive procedure.
4. Has symptoms for gastroparesis (GP) (that is, chronic postprandial fullness, abdominal pain, postprandial nausea, vomiting, loss of appetite and/or early satiety) the past 3 months.
5. Has documented slow gastric emptying (GE), with delayed GE by 13C-Spirulina gastric emptying breath test (GEBT) at Screening defined as >=80th percentile. Note: If a participant has had a documented scintigraphy or GEBT within the last 12 months that confirms the diagnosis of delayed GE, a screening GEBT would not be required.
6. Has nausea subscale (of American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary [ANMS-GCSI-DD]) symptom score >=2 at least 3 of 7 days during Screening.
7. Has haemoglobin A1c (HBA1c) less than (<) 10 percent (%) (for diabetes mellitus only).

Exclusion Criteria

The participant must be excluded from participating in the trial if the participant:

1. Has acute severe gastroenteritis and pronounced dehydration in the past 48 hours prior to Screening, gastric pacemaker, chronic parenteral feeding or persistent severe vomiting.
2. Has a known disturbance of small intestinal absorption, exocrine pancreatic function, liver metabolism, and pulmonary function.
3. Has a history of anorexia nervosa or bulimia.
4. Previous history of bezoars (the presence of retained liquid, bile, or small amounts of poorly organized food residue is permitted).
5. Difficulty swallowing solid food or pills.
6. Prior surgery involving the luminal gastrointestinal (GI) tract (cholecystectomy, appendectomy, and hysterectomy are permitted if performed greater than (>) 3 months prior to SmartPill test).
7. Any abdominal or pelvic surgery within the past 3 months.
8. Known or history of inflammatory bowel disease.
9. Has active diverticulitis, diverticular stricture, and other intestinal strictures.
10. Had major surgery, donated or lost 1 unit of blood (approximately 500 milliliter [mL]) within 4 weeks prior to the pretrial (screening) visit milligram per deciliter (mg/dL) (14.99 millimole per liter [mmol/L]) during any visit up to and including the randomization visit (Period 1 Day 1 predose). Note: If the participant meets this exclusion criterion and the investigator believes that the value is not consistent with the participant's current self-monitoring blood glucose values, the participant should not be excluded at this time. The visit can be repeated within 5 to 7 days.
11. Has had diabetic ketoacidosis (within the prior 4 weeks).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (9):
- United States (9):
  - 9171 West Thunderbird Road, Peoria, Arizona
  - 850 North Kolb Road, Tucson, Arizona
  - 11219 Financial Centre Parkway, Little Rock, Arkansas
  - 13055 Southwest 42nd Street, Miami, Florida
  - 8200 Southwest 117th Avenue, Miami, Florida
  - 125 Clairemont Avenue, Decatur, Georgia
  - 616 South Washington Street, Bastrop, Louisiana
  - 6035 Shallowford Road, Chattanooga, Tennessee
  - 26 Stonecreek Circle, Jackson, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Kuo B, Scimia C, Dukes G, Zhang W, Gupta S, Chen C, Chuang E, Camilleri M. Randomised clinical trial: safety, pharmacokinetics and pharmacodynamics of trazpiroben (TAK-906), a dopamine D2 /D3 receptor antagonist, in patients with gastroparesis. Aliment Pharmacol Ther. 2021 Aug;54(3):267-280. doi: 10.1111/apt.16451. Epub 2021 Jun 20. PMID 34148244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in the United States from 26 September 2017 to 09 March 2018.
Pre-assignment Details: Participants with a diagnosis of diabetes mellitus and gastroparesis (GP) or with idiopathic gastroparesis (IG) were enrolled. 51 participants were randomized in Part 1, out of which 48 completed the Part 1, 21 of 48 participants entered the Part 2.
Groups:
- Part 2: TAK-906 Maleate 25 mg Under Fed Conditions: TAK-906 maleate 1x25 mg, capsule, orally, once on Day 1 of Period 1 under fed (high fat breakfast) followed by fasted condition. There was a minimum 7- day washout period between the two conditions.
- Part 2: Metoclopramide 10 mg: Metaclopramide 10 mg, tablet, orally, once, 1 hour prior to breakfast on Day 1 in Part 2. There was a minimum 7- day washout period between the two conditions.
Period: Part 1 (Days 1 to 9)
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg | Part 2: TAK-906 Maleate 25 mg Under Fed Conditions | Part 2: TAK-906 Maleate 25 mg Fasted Condition | Part 2: Metoclopramide 10 mg
Started | 12 | 14 | 12 | 13 | 0 | 0 | 0
Completed | 11 | 14 | 12 | 11 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Days 17 to 25
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg | Part 2: TAK-906 Maleate 25 mg Under Fed Conditions | Part 2: TAK-906 Maleate 25 mg Fasted Condition | Part 2: Metoclopramide 10 mg
Started | 0 | 0 | 0 | 0 | 6 | 0 | 15
Treated | 0 | 0 | 0 | 0 | 6 | 0 | 13
Completed | 0 | 0 | 0 | 0 | 6 | 0 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Reason not specified | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Part 2: Period 2: Fasted (Day 25)
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg | Part 2: TAK-906 Maleate 25 mg Under Fed Conditions | Part 2: TAK-906 Maleate 25 mg Fasted Condition | Part 2: Metoclopramide 10 mg
Started | 0 | 0 | 0 | 0 | 0 | 6 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS), Part 1, included all participants who were randomized (Part 1) and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg | Total
Number analyzed (Participants) | 12 | 14 | 12 | 13 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (13.84) | 54.7 (11.75) | 52.7 (17.13) | 55.9 (10.19) | 53.4 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 10 | 10 | 40
  Male | 3 | 3 | 2 | 3 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 3 | 7 | 24
  Non-Hispanic and Latino | 3 | 9 | 9 | 6 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 1 | 4 | 2 | 8
  White | 11 | 13 | 7 | 11 | 42
  Multiracial | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 14 | 12 | 13 | 51
Height [Mean (Standard Deviation); unit: cm] | 164.62 (9.790) | 163.95 (6.751) | 164.56 (7.204) | 164.93 (9.778) | 164.50 (8.212)
Weight [Mean (Standard Deviation); unit: kg] | 74.70 (17.231) | 79.86 (13.470) | 80.55 (11.346) | 88.24 (11.803) | 80.95 (14.064)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight/[height^2]
  kg/m^2 | 27.282 (4.2276) | 29.679 (4.5043) | 29.832 (4.5461) | 32.565 (4.4001) | 29.887 (4.6805)
Underlying Disease [Count of Participants; unit: Participants]
  Diabetic Gastroparesis (DG) | 8 | 10 | 8 | 8 | 34
  Idiopathic Gastroparesis (IG) | 4 | 4 | 4 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced At Least One or More Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A SAE is an AE resulting in any of the following outcomes or deemed significant for any following reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event.
Time Frame: From Baseline to 14 days after the last dose of study drug (Up to approximately 39 days)
Population: SAS included all participants who were randomized (Part 1) or enrolled (Part 2) and received at least 1 dose of study drug in the respective part.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: TAK-906 Maleate 25 mg Fed Condition: TAK-906 maleate 1x25 mg, capsule, orally, once on Day 1 of Period 1 under fed (high fat breakfast) conditions followed by minimum 7- day washout period.
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg | Part 2: TAK-906 Maleate 25 mg Fed Condition | Part 2: TAK-906 Maleate 25 mg Fasted Condition | Part 2: Metoclopramide 10 mg
Number analyzed (Participants) | 12 | 14 | 12 | 13 | 6 | 6 | 13
Participants
  TEAEs | 4 | 4 | 3 | 4 | 1 | 0 | 1
  SAEs | 1 | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Markedly Abnormal Laboratory Parameters Values
Description: Clinical Laboratory parameters included tests for chemistry, hematology and urinalysis. Markedly abnormal values during treatment period were categorized as:alanine aminotransferase (ALT)>3.0 U/L*upper limit of normal(ULN),albumin<25 g/L*lower limit of normal(LLN),alkaline phosphatase >3.0 U/L*ULN,aspartate aminotransferase >3.0 U/L*ULN,bilirubin >2 umol/L*ULN,blood urea nitrogen(BUN) >10.7 mmol/L,calcium <1.75 mmol/L, >2.88 mmol/L,chloride <75 mmol/L, >126 mmol/L,creatinine >177umol/L,gamma glutamyl transferase (GGT) >3 U/L*ULN,glucose <2.8 mmol/L, >19.4 mmol/L,phosphate <0.52 mmol/L, >2.10 mmol/L,potassium<3 mmol/L, >6 mmol/L,sodium <130 mmol/L, >150 mmol/L,hematocrit (%) <0.8*LLN, >1.2*ULN,hemoglobin <0.8 g/L*LLN, >1.2 g/L*ULN,leukocytes <0.5 (10^9/L)*LLN, >1.5 (10^9/L)*ULN,erythrocytes<0.8 (10^12/L)*LLN, >1.2(10^12/L)*ULN,platelets <75(10^9/L), >600(10^9/L). Participants with at least 1 markedly abnormal laboratory parameter value is reported.
Time Frame: From Baseline to 14 days after the last dose of study drug in Part 1 (Up to approximately 23 days)
Population: SAS included all participants who were randomized and received at least 1 dose of study drug in the Part 1. Laboratory assessment were performed only in Part 1 of the study. Number analyzed are participants with data available for the particular parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg
Number analyzed (Participants) | 12 | 14 | 12 | 13
Participants
  Hematocrit (%)<0.8 x LLN: number analyzed (Participants) | 12 | 13 | 12 | 12
  Hematocrit (%)<0.8 x LLN | 0 | 1 | 0 | 0
  Hemoglobin (g/L) <0.8 x LLN: number analyzed (Participants) | 12 | 13 | 12 | 12
  Hemoglobin (g/L) <0.8 x LLN | 1 | 0 | 0 | 0
  ALT >3.0 U/Lx ULN: number analyzed (Participants) | 12 | 13 | 12 | 12
  ALT >3.0 U/Lx ULN | 0 | 0 | 1 | 0
  AST >3.0 U/L x ULN: number analyzed (Participants) | 12 | 13 | 12 | 12
  AST >3.0 U/L x ULN | 0 | 0 | 1 | 0
  BUN >10.7 mmol/L: number analyzed (Participants) | 12 | 13 | 12 | 12
  BUN >10.7 mmol/L | 1 | 0 | 0 | 1
  Calcium >2.88 mmol/L: number analyzed (Participants) | 12 | 13 | 12 | 12
  Calcium >2.88 mmol/L | 0 | 0 | 0 | 1
  GGT >3 x ULN: number analyzed (Participants) | 12 | 10 | 11 | 12
  GGT >3 x ULN | 0 | 0 | 0 | 1
  Sodium (mmol/L) <130 mmol/L: number analyzed (Participants) | 12 | 13 | 12 | 12
  Sodium (mmol/L) <130 mmol/L | 1 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Markedly Abnormal Vital Signs
Description: Vital signs included body temperature, diastolic and systolic blood pressure (mmHg), and heart rate (beats per minute [bpm]). Heart rate<50 bpm and systolic blood pressure <85 mmHg were considered markedly abnormal.
Time Frame: From Baseline to 14 days after the last dose of study drug (Up to approximately 39 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg | Part 2: TAK-906 Maleate 25 mg Fed Condition | Part 2: TAK-906 Maleate 25 mg Fasted Condition | Part 2: Metoclopramide 10 mg
Number analyzed (Participants) | 12 | 14 | 12 | 13 | 6 | 6 | 13
Participants
  Heart Rate (bpm) <50 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure (mmHg) <85 | 1 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Markedly Abnormal Electrocardiogram (ECG) Values
Description: The 12-lead electrocardiogram (ECG) values outside the range Heart Rate <50 (beats/min), PR Interval ≤120 (msec), PR Interval ≥200 (msec), QRS Duration ≥120 (msec), QT Interval ≥460 (msec) were considered markedly abnormal.
Time Frame: From Baseline to 14 days after the last dose of study drug (Up to approximately 39 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg | Part 2: TAK-906 Maleate 25 mg Fed Condition | Part 2: TAK-906 Maleate 25 mg Fasted Condition | Part 2: Metoclopramide 10 mg
Number analyzed (Participants) | 12 | 14 | 12 | 13 | 6 | 6 | 13
Participants
  Heart Rate (bpm) <50 | 1 | 1 | 0 | 0 | 1 | 1 | 0
  PR Interval (msec) ≤120 | 0 | 1 | 1 | 1 | 0 | 0 | 1
  PR Interval (msec) ≥200 | 1 | 2 | 1 | 4 | 0 | 0 | 4
  QRS Duration (msec) ≥120 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  QT Interval (msec) ≥460 | 0 | 1 | 0 | 1 | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Serum Prolactin Concentration on Day 1 at Tmax, Time of First Occurrence of Maximum Serum Concentration (Cmax) for TAK-906 Maleate for Part 1
Description: Change in serum prolactin on Day 1 at the Tmax, time of first occurrence of maximum serum concentration (Cmax) relative to Baseline was calculated as a ratio of maximum serum prolactin concentration on Day 1 to serum prolactin concentration at Baseline.
Time Frame: Day 1 predose (Baseline), 1 hour and at multiple timepoints (Up to 8 hours) postdose
Population: Full analysis set (FAS) included all participants who were randomized (Part 1), received at least 1 dose of study drug, had a baseline value, and had at least 1 valid postbaseline value for at least one of pharmacodynamic (PD) measurement. Overall number of participants analyzed are participants with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg
Number analyzed (Participants) | 12 | 14 | 11 | 13
ratio | 1.54 (0.704) | 12.77 (9.102) | 19.92 (13.604) | 20.07 (9.170)
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 5 mg; Change in serum prolactin on Day 1 at the Tmax as a ratio of Cmax to serum prolactin concentration at Baseline; Test type: Other; p < 0.001, ANCOVA — ANCOVA model was used for analysis. Treatment, underlying disease (DG/IG) were fixed factors. ln of baseline prolactin concentration as covariate, ln of ratio of Cmax to baseline concentration as response. Results in original scale are presented; Least Square (LS) Mean Difference = 7.38, 95% CI 2-sided [4.03 to 13.52]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 25 mg; Change in serum prolactin on Day 1 at the Tmax as a ratio of Cmax to serum prolactin concentration at Baseline; Test type: Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 11.24, 95% CI 2-sided [5.91 to 21.41]
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 100 mg; Change in serum prolactin on Day 1 at the Tmax as a ratio of Cmax to serum prolactin concentration at Baseline; Test type: Other; p < 0.001, ANCOVA — ANCOVA model was used for analysis. Treatment, underlying disease (DG/IG) were fixed factors. ln of baseline prolactin concentration - covariate, ln of ratio of Cmax to baseline concentration as response. Results in original scale are presented; LS Mean Difference = 12.80, 95% CI 2-sided [6.94 to 23.59]

6. Secondary Outcome: Change From Baseline in Gastric Emptying Breath Test (GEBT) Gastric Half-emptying Time as Measured by the 13C Spirulina GEBT Following Multiple Dose Administration of TAK-906 Maleate on Day 7 for Part 1
Description: The GEBT is a nonradioactive, noninvasive, orally administered test for measuring the rate of solid phase gastric emptying (GE) in adults. The GEBT measures how fast solid food moves from the stomach to the small intestine during the digestive process and aids in the diagnosis of delayed stomach emptying (GP). GE half-emptying time is the time in minutes (min) for half of the ingested solids to leave the stomach. This value was measured by the 13C spirulina GEBT.
Time Frame: Baseline and Day 7
Population: FAS included all participants who were randomized (Part 1), received at least 1 dose of study drug, had a baseline value, and had at least 1 valid postbaseline value for assessment of at least one of the PD measurement. Overall number of participants analyzed are the participants with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg
Number analyzed (Participants) | 11 | 14 | 11 | 13
min
  Baseline | 118.74 (43.106) | 130.18 (35.316) | 121.26 (33.606) | 122.50 (31.803)
  Change from Baseline at Day 7: number analyzed (Participants) | 10 | 14 | 10 | 10
  Change from Baseline at Day 7 | 4.55 (16.332) | 6.21 (36.986) | 7.80 (52.946) | 7.72 (24.609)
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 5 mg; Change from Baseline in GEBT gastric half-emptying time on Day 7 in Part 1; Test type: Other; p = 0.599, ANCOVA — P-value was obtained by ANCOVA model with treatment and underlying disease (DG/IG) condition as fixed factors and baseline score as covariate; LS Mean Difference = 7.76, 95% CI 2-sided [-21.89 to 37.41], Standard Error of Mean 14.648
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 25 mg; Change from Baseline in GEBT gastric half-emptying time on Day 7 in Part 1; Test type: Other; p = 0.687, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 6.28, 95% CI 2-sided [-25.04 to 37.59], Standard Error of Mean 15.469
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 100 mg; Change from Baseline in GEBT gastric half-emptying time on Day 7 in Part 1; Test type: Other; p = 0.605, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 8.05, 95% CI 2-sided [-23.22 to 39.33], Standard Error of Mean 15.450

7. Secondary Outcome: Change From Baseline in Gastric Emptying Breath Test (GEBT) Gastric Half-emptying Time Following Single Dose Administration of TAK-906 Maleate as Measured by the 13C Spirulina GEBT on Day 1
Description: as for outcome 6
Time Frame: Baseline and Day 1 of Part 1
Population: FAS included all participants who were randomized (Part 1), received at least 1 dose of study drug, had a baseline at least 1 valid postbaseline value for assessment of at least one PD measurement. Overall number of participants analyzed are participants with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: minute (min)
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg
Number analyzed (Participants) | 11 | 14 | 11 | 13
minute (min)
  Baseline | 118.74 (43.106) | 130.18 (35.316) | 121.26 (33.606) | 122.50 (31.803)
  Change from Baseline at Day 1: number analyzed (Participants) | 11 | 13 | 11 | 13
  Change from Baseline at Day 1 | -5.71 (21.687) | 0.12 (21.736) | 6.74 (44.390) | 0.71 (21.192)
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 5 mg; Change from Baseline in GEBT gastric half-emptying time on Day 1 in Part 1; Test type: Other; p = 0.522, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 7.56, 95% CI 2-sided [-16.06 to 31.19], Standard Error of Mean 11.708
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 25 mg; Change from Baseline in GEBT gastric half-emptying time on Day 1 in Part 1; Test type: Other; p = 0.293, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 12.92, 95% CI 2-sided [-11.58 to 37.43], Standard Error of Mean 12.143
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 100 mg; Change from Baseline in GEBT gastric half-emptying time on Day 1 in Part 1; Test type: Other; p = 0.551, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 7.00, 95% CI 2-sided [-16.52 to 30.52], Standard Error of Mean 11.654

8. Secondary Outcome: Percent Change From Baseline in Gastric Emptying (GE) Time as Measured by the SmartPill on Day 7 for Part 1
Description: SmartPill is an ingestible capsule that measures pressure, potential of hydrogen (pH) and temperature as it travels through the gastrointestinal (GI) tract to assess GE and GI motility. SmartPill eliminates radiation exposure and is the only motility test that provides a complete transit profile of the GI tract.
Time Frame: Baseline and Day 7
Population: FAS included all participants who were randomized (Part 1), received at least 1 dose of study drug, had a baseline value, and had at least 1 valid postbaseline value for assessment of at least one of the PD measurements. Overall number of participants analyzed is number of participants with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change in GE time
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg
Number analyzed (Participants) | 8 | 10 | 9 | 8
percent change in GE time | 124.62 (181.125) | 61.72 (195.867) | 419.27 (885.362) | 71.09 (121.584)
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 5 mg; Percent Change in GE time measured by the SmartPill on Day 7 in Part 1; Test type: Other; p = 0.274, Wilcoxon Rank Sum tests — P-value was obtained with pairwise Wilcoxon Rank Sum tests; Hodges-Lehmann Estimate of Median Diff = -18.14, 95% CI 2-sided [-307.58 to 13.56]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 25 mg; Percent Change in GE time measured by the SmartPill on Day 7 in Part 1; Test type: Other; p = 0.481, Wilcoxon Rank Sum tests — P-value was obtained with pairwise Wilcoxon Rank Sum tests; Hodges-Lehmann Estimate of Median Diff = -26.95, 95% CI 2-sided [-229.73 to 530.49]
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1: TAK 906 Maleate 100 mg; Percent Change in GE on time measured by the SmartPill Day 7 in Part 1; Test type: Other; p = 0.382, Wilcoxon Rank Sum tests — P-value was obtained with pairwise Wilcoxon Rank Sum tests; Hodges-Lehmann Estimate of Median Diff = -24.49, 95% CI 2-sided [-225.87 to 98.91]

9. Secondary Outcome: AUCτ: Area Under the Plasma Concentration-time Curve From 0 to Time (T) Over the Dosing Interval for TAK-906 in Part 1
Time Frame: Part 1: Day 1 predose and at multiple timepoints, (Up to 8 hours) postdose and Day 7 predose and at multiple timepoints (Up to 48 hours) postdose
Population: Pharmacokinetic (PK) set included participants who were randomized and received at least 1 dose of study drug and had at least 1 measurable plasma TAK-906 concentration. Overall number of participants analyzed are participants with data available for analysis of AUCt. Number analyzed are participants with evaluable data at given time-point.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg
Number analyzed (Participants) | 13 | 11 | 12
h*ng/mL
  Day 1: number analyzed (Participants) | 12 | 11 | 12
  Day 1 | 4.67 (1.69) | 23.0 (7.76) | 131 (44.8)
  Day 7: number analyzed (Participants) | 13 | 11 | 10
  Day 7 | 5.46 (2.07) | 26.3 (11.3) | 166 (93.0)

10. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK 906 in Part 1
Time Frame: as for outcome 9
Population: PK set included participants who were randomized and received at least 1 dose of study drug and had at least 1 measurable plasma TAK-906 concentration. Overall number of participants analyzed are participants with data available for analysis of Cmax. Number analyzed are participants with evaluable data at given time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg
Number analyzed (Participants) | 13 | 11 | 13
ng/mL
  Day 1: number analyzed (Participants) | 12 | 11 | 13
  Day 1 | 2.27 (0.819) | 12.0 (5.36) | 75.7 (39.9)
  Day 7: number analyzed (Participants) | 13 | 11 | 10
  Day 7 | 2.87 (1.78) | 15.5 (5.58) | 99.6 (69.4)

11. Secondary Outcome: Ctrough: Observed Concentration at the End of a Dosing Interval for TAK-906 in Part 1
Time Frame: Part 1: Predose on Days 2, 3, 4, 5, 6, 7, 8 and 9
Population: PK set included participants who were randomized and received at least 1 dose of study drug and had at least 1 measurable plasma TAK-906 concentration. Overall number of participants analyzed are participants with data available for analysis of Ctrough. Number analyzed are participants with evaluable data at given time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg
Number analyzed (Participants) | 13 | 11 | 13
ng/mL
  Predose on Day 2: number analyzed (Participants) | 13 | 10 | 13
  Predose on Day 2 | 0.0121 (0.0315) | 0.262 (0.349) | 0.770 (0.513)
  Predose on Day 3: number analyzed (Participants) | 13 | 10 | 12
  Predose on Day 3 | 0.0423 (0.0527) | 0.503 (0.640) | 0.958 (0.750)
  Predose on Day 4: number analyzed (Participants) | 13 | 11 | 12
  Predose on Day 4 | 0.0178 (0.0503) | 0.302 (0.214) | 1.17 (0.799)
  Predose on Day 5: number analyzed (Participants) | 13 | 11 | 11
  Predose on Day 5 | 0.0457 (0.0962) | 1.09 (1.97) | 1.95 (2.38)
  Predose on Day 6: number analyzed (Participants) | 11 | 11 | 11
  Predose on Day 6 | 0.0423 (0.0502) | 0.412 (0.415) | 1.01 (0.469)
  Predose on Day 7: number analyzed (Participants) | 13 | 11 | 10
  Predose on Day 7 | 0.0596 (0.0905) | 0.336 (0.383) | 1.48 (0.936)
  Predose on Day 8: number analyzed (Participants) | 13 | 11 | 11
  Predose on Day 8 | 0.0763 (0.100) | 0.522 (0.648) | 1.16 (0.878)
  Predose on Day 9: number analyzed (Participants) | 13 | 11 | 10
  Predose on Day 9 | 0.0700 (0.120) | 0.280 (0.243) | 1.40 (1.08)

12. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-906 in Part 1
Time Frame: as for outcome 9
Population: PK set included participants who were randomized and received at least 1 dose of study drug and had at least 1 measurable plasma TAK-906 concentration. Overall number of participants analyzed are participants with data available for analysis of Tmax. Number analyzed are participants with evaluable data at given time-point.
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg
Number analyzed (Participants) | 13 | 11 | 13
hour (hr)
  Day 1: number analyzed (Participants) | 12 | 11 | 13
  Day 1 | 1.00 [0.48 to 2.00] | 1.00 [0.50 to 4.00] | 1.00 [0.50 to 2.00]
  Day 7: number analyzed (Participants) | 13 | 11 | 10
  Day 7 | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 1.52] | 0.98 [0.48 to 1.98]

ADVERSE EVENTS:
Time Frame: Baseline to 14 days after the last dose of study drug (Up to approximately 39 days)
Description: Collection of AEs was commenced at the time the subject signed the informed consent and continued until 14 days after the last dose of investigational product. At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1: Placebo | Part 1: TAK 906 Maleate 5 mg | Part 1: TAK 906 Maleate 25 mg | Part 1: TAK 906 Maleate 100 mg | Part 2: TAK-906 Maleate 25 mg Fed Condition | Part 2: TAK-906 Maleate 25 mg Fasted Condition | Part 2: Metoclopramide 10 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/12 | 0/13 | 0/6 | 0/6 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/14 | 0/12 | 1/13 | 0/6 | 0/6 | 0/13
Other Adverse Events (participants affected / at risk) | 3/12 | 4/14 | 3/12 | 4/13 | 1/6 | 0/6 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=12) | Part 1: TAK 906 Maleate 5 mg (N=14) | Part 1: TAK 906 Maleate 25 mg (N=12) | Part 1: TAK 906 Maleate 100 mg (N=13) | Part 2: TAK-906 Maleate 25 mg Fed Condition (N=6) | Part 2: TAK-906 Maleate 25 mg Fasted Condition (N=6) | Part 2: Metoclopramide 10 mg (N=13)
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=12) | Part 1: TAK 906 Maleate 5 mg (N=14) | Part 1: TAK 906 Maleate 25 mg (N=12) | Part 1: TAK 906 Maleate 100 mg (N=13) | Part 2: TAK-906 Maleate 25 mg Fed Condition (N=6) | Part 2: TAK-906 Maleate 25 mg Fasted Condition (N=6) | Part 2: Metoclopramide 10 mg (N=13)
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 — Participant in Part 1: TAK 906 Maleate 100 mg had an AE of liver function test increased on Day 1. The blood draw for the liver function tests was done prior to the first study drug administration.
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — A mild AE of tremor occurred in 1 participant (had history of diabetes) in Part 1:TAK 906 Maleate 100 mg arm, on Day 3, resolved on Day 4, considered not related by investigator. No other signs/symptoms of neurological origin were observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03268941/SAP_000.pdf
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03268941/Prot_001.pdf